CLINICAL TRIAL: NCT00288067
Title: A Phase I-II Trial of Fenretinide (4-HPR) + Rituximab in Patients With B-cell Lymphoma
Brief Title: Fenretinide and Rituximab in Treating Patients With B-Cell Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: NCI stopped supplying fenretinide in November of 2012.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00104; NCI-2009-00104 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000456502 (Other: NCI); UWCC-UW-6071 (Other: Fred Hutchinson Cancer Research Center); UWCC-06-0644-H/A (Other: Fred Hutchinson Cancer Research Center); UWCC-6071 (Other: Fred Hutchinson Cancer Research Center); FHCRC-6071 (Other: Fred Hutchinson Cancer Research Center); 6071 (Other: University of Washington Medical Center); 6957 (Other: CTEP); R21CA119519 (NIH)
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-01

CONDITIONS: Adult Nodular Lymphocyte Predominant Hodgkin Lymphoma; B-cell Chronic Lymphocytic Leukemia; Contiguous Stage II Adult Burkitt Lymphoma; Contiguous Stage II Adult Diffuse Large Cell Lymphoma; Contiguous Stage II Adult Lymphoblastic Lymphoma; Contiguous Stage II Grade 1 Follicular Lymphoma; Contiguous Stage II Grade 2 Follicular Lymphoma; Contiguous Stage II Mantle Cell Lymphoma; Stage II Marginal Zone Lymphoma; Stage II Small Lymphocytic Lymphoma; Extranodal Marginal Zone B-cell Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Noncontiguous Stage II Adult Burkitt Lymphoma; Noncontiguous Stage II Adult Diffuse Large Cell Lymphoma; Noncontiguous Stage II Adult Lymphoblastic Lymphoma; Noncontiguous Stage II Grade 1 Follicular Lymphoma; Noncontiguous Stage II Grade 2 Follicular Lymphoma; Noncontiguous Stage II Mantle Cell Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Splenic Marginal Zone Lymphoma; Stage I Adult Burkitt Lymphoma; Stage I Adult Diffuse Large Cell Lymphoma; Stage I Adult Hodgkin Lymphoma; Stage I Adult Lymphoblastic Lymphoma; Stage I Chronic Lymphocytic Leukemia; Stage I Grade 1 Follicular Lymphoma; Stage I Grade 2 Follicular Lymphoma; Stage I Small Lymphocytic Lymphoma; Stage II Adult Hodgkin Lymphoma; Stage II Chronic Lymphocytic Leukemia; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Hodgkin Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Chronic Lymphocytic Leukemia; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Small Lymphocytic Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Chronic Lymphocytic Leukemia; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Small Lymphocytic Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Hodgkin Disease; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Waldenstrom Macroglobulinemia | interventions — Fenretinide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (fenretinide, rituximab) (Experimental): PHASE I: Patients receive fenretinide PO BID on days 1-5. Treatment repeats weekly for at least 4 weeks in the absence of disease progression or unacceptable toxicity.
  PHASE II: Patients receive fenretinide PO BID on days 1-5 in weeks 1-8 and rituximab IV once weekly in weeks 5-8. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: fenretinide; Drug: rituximab

INTERVENTIONS:
Drug: fenretinide — Given PO
  Other Names: fenretinimide; McN-R-1967
Drug: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan

SUMMARY:
This phase I/II trial is studying the side effects and best dose of fenretinide and to see how well it works when given together with rituximab in treating patients with B-cell non-Hodgkin lymphoma. Drugs used in chemotherapy, such as fenretinide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some find cancer cells and kill them or carry cancer-killing substances to them. Others interfere with the ability of cancer cells to grow and spread. Giving fenretinide together with rituximab may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety of fenretinide delivered in a 5 of 7 day regimen. (Phase I) II. To estimate the efficacy (response rates) of fenretinide + rituximab in patients with B-cell non-Hodgkin lymphoma (NHL). (Phase II)

SECONDARY OBJECTIVES:

I. To perform pharmacokinetic studies on patients receiving fenretinide. (Phase I) II. To determine the intratumoral concentrations of fenretinide. (Phase I) III. To evaluate the in vivo mechanism of action of fenretinide. (Phase I) IV. To identify the predictors of response to fenretinide. (Phase I) V. To estimate the response rates, positron emission tomography (PET) response, overall survival (OS), progression-free survival (PFS), time to progression (TTP), and disease-free survival (DFS) of patients treated on this study. (Phase I) VI. To estimate the overall survival (OS), progression-free survival (PFS), time to progression (TTP), disease-free survival (DFS), and PET responses of patients treated on this study. (Phase II) VII. To perform pharmacokinetic studies on patients receiving fenretinide. (Phase II) VIII. To determine the intratumoral concentration of fenretinide. (Phase II) IX. To identify the predictors of response to fenretinide and fenretinide + rituximab in B-NHL. (Phase II) X. To evaluate the in vivo mechanism of action of fenretinide in B-NHL. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of fenretinide followed by a phase II study.

PHASE I: Patients receive fenretinide orally (PO) twice daily (BID) on days 1-5. Treatment repeats weekly for at least 4 weeks in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients receive fenretinide PO BID on days 1-5 in weeks 1-8 and rituximab intravenously (IV) once weekly in weeks 5-8. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a confirmed cluster of differentiation (CD) 20+ lymphoid malignancy

  * All patients with indolent NHL (including Follicular, Marginal Zone, small lymphocytic lymphoma (SLL)/chronic lymphocytic leukemia (CLL), lymphoplasmacytoid/Waldenström's, nodular lymphocyte predominant Hodgkins) are potentially eligible
  * Patients with Aggressive Lymphoma (including diffuse large B-cell, Burkitt's, Burkitt's-like, B-lymphoblastic) may be considered for this protocol only if unable or unwilling to receive potentially curative intensive therapy
  * All Mantle Cell Lymphoma patients are potentially eligible
* The World Health Organization (WHO) classification of patient's malignancy must be provided
* Patients must have a Southwest Oncology Group (SWOG)/Eastern Cooperative Oncology Group (ECOG) of =< 2
* Patients should have an expected survival if untreated of at least 60 days
* Patients must be expected to complete at least 8 weeks of therapy
* Serum bilirubin less than 2 times the upper limit of normal and no other serious medical condition
* Creatinine less than 2 times the upper limit of normal and no other serious medical condition
* Patients must have measurable disease defined as lesions that can be accurately measured in two dimensions by computed tomography (CT), magnetic resonance imaging (MRI), medical photograph (skin or oral lesion), plain x-ray, or other conventional technique and a greatest transverse diameter of 1 cm or greater; or palpable lesions with both diameters >= 2 cm or evaluable disease in the bone marrow; patients must have a CT of chest, abdomen, and pelvis within 28 days of enrollment; patients with evidence of adenopathy in the neck must have a CT of the neck; (Note: Patients with CLL do not need to have radiographically measurable disease as this is not required to measure response in this disease setting)
* All patients with an unknown prior bone marrow status or history of bone marrow involvement must have a bone marrow aspirate and biopsy within 28 days of enrollment and no intervening anticancer therapy
* All patients must be informed of the investigational nature of this study and have given written consent in accordance with institutional and federal guidelines

Exclusion Criteria:

* Patients known to be human immunodeficiency virus (HIV) positive
* Patients with evidence of active central nervous system malignancy
* Pregnant or nursing women
* Men or women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method
* Concurrent anti-neoplastic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2005-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Gopal, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Fenretinide and Rituximab: PHASE I: Patients receive fenretinide PO BID on days 1-5. Treatment repeats weekly for at least 4 weeks in the absence of disease progression or unacceptable toxicity.
  PHASE II: Patients receive fenretinide PO BID on days 1-5 in weeks 1-8 and rituximab IV once weekly in weeks 5-8. Treatment continues in the absence of disease progression or unacceptable toxicity.
  pharmacological study : Correlative studies
  rituximab : Given IV
  fenretinide : Given PO
Period: Overall Study
Arm/Group | Fenretinide and Rituximab
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fenretinide and Rituximab
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 26
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Safety, in Terms of Dose-limiting Toxicity (DLT) of 2 Daily Doses of Single Agent Fenretinide (Phase I)
Description: A group of 3 patients would start treatment ast the dose of 900mg/m^2 BID, and if none of the 3 experienced a DLT, another 3 would then be treated at that dose. Dose Limiting Toxicity was defined as any related toxicity of grade 4 or 5 on or before the completion of 4 weeks of therapy.
  Per response evaluation criteria 1999 Cheson Response Criteria for Malignant Lymphoma (CHESON99) for target lesions assessed by either CT or MRI:
  Complete Response (CR): Complete disappearance of all measurable and non-measurable disease; Complete Response Unconfirmed (CRU): Complete disappearance of all measurable and non-measurable disease, with the exception of all residual nodal masses >1.5cm in Greatest Transverse Diameter (GTD) reduced by 75% in Sum of the Product of the greatest Diameters (SPD); Partial Response (PR): 50% decrease in the SPD.
Time Frame: Number of participants that experienced a dose-limiting toxicity
Population: 7 participants were analyzed in the Rituximab Naive arm and 16 participants were analyzed in the Rituximab Pre Treated Arm.
Measure: Number; unit: participants
Arm/Group | Fenretinide and Rituximab
Number analyzed (Participants) | 23
participants | 0

2. Primary Outcome: Response Rates of B-Non-Hodgkin Lymphoma to the Combination of Rituximab and Fenretinide (Phase II)
Description: The trial was stratified into rituximab-naïve and rituximab pre-treated patients, and the target response rates for these groups were expected to be 30% and 10%, respectively. The numbers reported below are subjects who achieved a response of partial response or better.
Time Frame: Up to 7 years
Population: No subjects in Phase 1 met the DLT, therefore Phase II was conducted at 900mg/m2. Of the 32 subjects, 4 subjects were not evaluable for disease response (2 subjects in Phase 1 and 2 subjects in Phase 2).
Measure: Number; unit: participants
Groups:
- Fenretinide and Rituximab (Rituximab Naive); Fenretinide and Rituximab (Rituximab Pre Treated): PHASE II: Patients receive fenretinide PO BID on days 1-5 in weeks 1-8 and rituximab IV once weekly in weeks 5-8.
Arm/Group | Fenretinide and Rituximab (Rituximab Naive) | Fenretinide and Rituximab (Rituximab Pre Treated)
Number analyzed (Participants) | 7 | 16
participants | 4 | 0

ADVERSE EVENTS:
Arm/Group | Fenretinide and Rituximab
Serious Adverse Events (participants affected / at risk) | 6/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fenretinide and Rituximab (N=32)
Allergic Reaction (Immune system disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Infections and infestations - Other, specify, Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10 (Infections and infestations) | 1 (1)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify, Papillary Thy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fenretinide and Rituximab (N=32)
Night Blindness (Eye disorders) | 18 (53)
Abdominal Distention (Gastrointestinal disorders) | 2 (3)
Abdominal Pain (Gastrointestinal disorders) | 7 (16)
Alanine aminotransferase increased (Investigations) | 3 (3)
Alkaline phosphatase increased (Investigations) | 2 (3)
Allergic Reaction (Immune system disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 10 (22)
Anorexia (Metabolism and nutrition disorders) | 7 (7)
Anxiety (Psychiatric disorders) | 2 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 5 (8)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Blood Bilirubin Increased (Investigations) | 5 (7)
Blurred Vision (Eye disorders) | 4 (7)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 5 (11)
Bone Pain (Musculoskeletal and connective tissue disorders) | 3 (5)
Bruising (Injury, poisoning and procedural complications) | 2 (3)
Cataract (Eye disorders) | 3 (8)
Chills (General disorders) | 2 (2)
Cholesterol High (Investigations) | 2 (2)
Constipation (Gastrointestinal disorders) | 6 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (8)
Creatinine Increased (Investigations) | 7 (22)
Cytokine release syndrome (Immune system disorders) | 7 (18)
Depression (Psychiatric disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 12 (20)
Dizziness (Nervous system disorders) | 7 (7)
Dry Eye (Eye disorders) | 5 (7)
Dry Skin (Skin and subcutaneous tissue disorders) | 9 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Edema Limbs (General disorders) | 6 (9)
Eye disorders - Other, specify, yellowing/discoloration of lights (Eye disorders) | 15 (17)
Eye disorders - Other, specify, Altered color perception (Eye disorders) | 4 (13)
Fatigue (General disorders) | 11 (33)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Fever (General disorders) | 2 (2)
Flashing Lights (Eye disorders) | 4 (4)
Flatulance (Gastrointestinal disorders) | 3 (4)
Fracture (Injury, poisoning and procedural complications) | 4 (6)
Hot Flashes (Vascular disorders) | 6 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (16)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (5)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 11 (21)
Hypocalcemia (Metabolism and nutrition disorders) | 16 (31)
Hypokalemia (Metabolism and nutrition disorders) | 5 (12)
Hyponatremia (Metabolism and nutrition disorders) | 6 (7)
Hypotension (Vascular disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 5 (5)
Lymphocyte Count Decreased (Investigations) | 9 (31)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5)
Nausea (Gastrointestinal disorders) | 3 (4)
Neutrophil Count Decreased (Investigations) | 9 (16)
Pain (General disorders) | 2 (2)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Peripheral Sensory Neuropathy (Nervous system disorders) | 6 (8)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Photosensitivity (Skin and subcutaneous tissue disorders) | 9 (20)
Platelet Count Decreased (Investigations) | 10 (29)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 20 (22)
Sinusitis (Infections and infestations) | 4 (4)
Thromboembolic Event (Vascular disorders) | 2 (2)
Upper Respiratory Infection (Infections and infestations) | 4 (4)
Urinary Frequency (Renal and urinary disorders) | 3 (4)
Urinary Tract Infection (Infections and infestations) | 2 (3)
Vaginal Infection (Infections and infestations) | 2 (3)
White Blood Cell Decreased (Investigations) | 9 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less